CLINICAL TRIAL: NCT02474914
Title: Efficacy of Octreotide in the Prevention of Postoperative Complications After Pancreaticodudenectomy in Patients With Soft Pancreas and Non-dilated Pancreatic Duct: A Prospective Randomized Trial"
Brief Title: Octreotide in the Prevention of Postoperative Complications After Pancreaticoduodenectomy
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Gastroenterology surgical center, mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Octreotide PD
Record Dates: First submitted 2015-06-13; First posted 2015-06-18 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2014-06

CONDITIONS: Periampullary Carcinoma Resectable
MeSH Terms: interventions — Octreotide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Octreotide (Active Comparator): Enrolled patients will be randomized to either the octreotide (sandostatin ) or the placebo group. The randomization process will be done using closed envelop method and will be withdrawn by a nurse after pancreaticoduodenectomy . Patients in the octreotide group will receive sandostatin 100ug SC every 8 hours daily staring from the day of operation to the postoperative day 7. Patients in the placebo group will receive saline administered in a similar manner.
  Interventions: Drug: Octreotide
- Placebo (Placebo Comparator): pancreaticoduodenectomy without octreotide postoperative
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octreotide — Octreotide will be given after PD
  Other Names: sandostatin
  Arms: Octreotide
Drug: Placebo — Octreotide will NOT be given after PD
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
pancreaticoduodenectomy (PD) is the standard operation for treatment of patients with benign and malignant pancreatic and periampullary diseases. Despite improved surgical technique and postoperative care, the mortality rate after PD is high reaching up to 30%, due to high incidence of postoperative complications . Pancreatic fistula (PF) is the one of the most frequent complications of PD and the major contributor to postoperative morbidity The aim of this study to evaluate the effect of the perioperative octreotide use after PD for prevention of the postoperative pancreatic fistula. The secondary outcomes are overall postoperative complications, mortality and the cost benefit relationship of the use of the perioperative octreotide.

DETAILED DESCRIPTION:
This study will be a prospective randomized controlled trial for perioperative use of octreotide in patients after PD for pancreatic and periampullary tumours from May 2014 to April 2017 in Gastroenterology surgical center, Mansoura University, Egypt.

The primary outcome of the study is the effect of perioperative use of octreotide on the rate of development of postoperative pancreatic fistula in patients after PD for pancreatic and periampullary tumours. The secondary outcome is postoperative overall complications, mortality, duration of the hospital length of stay and cost-benefit relationship of perioperative use of octreotide.

Enrolled patients will be randomized to either the octreotide or the placebo group. The randomization process will be done using closed envelop method and will be withdrawn by a nurse after pancreaticoduodenectomy . Patients in the octreotide group will receive sandostatin 100ug SC every 8 hours daily staring from the day of operation to the postoperative day 7. Patients in the placebo group will receive saline administered in a similar manner.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with pancreatic and periampullary tumours anticipated for PD will be eligible to participate in this trial.
2. patients with non dilated pancreatic duct and soft pancreas

Exclusion Criteria:

Exclusion criteria:

1. Age over 70.
2. Patients who underwent total or distal pancreatic resection.
3. Patients with unresectable disease who will undergo any surgical procedure other than PD for pancreatic and periampullary tumours.
4. Patients underwent neoadjuvant chemotherapy or radiotherapy.
5. PD more than 3mm.
6. firm pancreas.
7. PJ

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
the rate of development of postoperative pancreatic fistula | 30 day
  POPF was defined by International Study Group of Pancreatic Fistula (ISGPF) as any volume of drained fluid on or after postoperative day (POD) 3 with amylase content greater than 3 times the serum amylase activity . POPF was graded into Grade A, B, and C according to the clinical course

SECONDARY OUTCOMES:
Delayed gastric emptying | 30 days
  Delayed gastric emptying was defined as output from a nasogastric tube of greater than 500 ml per day that persisted beyond 10th POD, the failure to maintain oral intake by 14th POD, or reinsertion of a nasogastric tube. Biliary leak was defined as the presence of bile in the drainage fluid that persists to 4th POD
duration of the hospital length of stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Principal Investigator — Mansoura University
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Mansoura, Egypt

REFERENCES:
- [Background] Lowy AM, Lee JE, Pisters PW, Davidson BS, Fenoglio CJ, Stanford P, Jinnah R, Evans DB. Prospective, randomized trial of octreotide to prevent pancreatic fistula after pancreaticoduodenectomy for malignant disease. Ann Surg. 1997 Nov;226(5):632-41. doi: 10.1097/00000658-199711000-00008. PMID 9389397
- [Result] El Nakeeb A, Salah T, Sultan A, El Hemaly M, Askr W, Ezzat H, Hamdy E, Atef E, El Hanafy E, El-Geidie A, Abdel Wahab M, Abdallah T. Pancreatic anastomotic leakage after pancreaticoduodenectomy. Risk factors, clinical predictors, and management (single center experience). World J Surg. 2013 Jun;37(6):1405-18. doi: 10.1007/s00268-013-1998-5. PMID 23494109
- [Result] Penumadu P, Barreto SG, Goel M, Shrikhande SV. Pancreatoduodenectomy - preventing complications. Indian J Surg Oncol. 2015 Mar;6(1):6-15. doi: 10.1007/s13193-013-0286-z. Epub 2014 Jan 19. PMID 25937757
- [Result] Hashimoto D, Chikamoto A, Ohmuraya M, Hirota M, Baba H. Pancreaticodigestive anastomosis and the postoperative management strategies to prevent postoperative pancreatic fistula formation after pancreaticoduodenectomy. Surg Today. 2014 Jul;44(7):1207-13. doi: 10.1007/s00595-013-0662-x. Epub 2013 Jul 11. PMID 23842691
- [Result] Fernandez-Cruz L, Jimenez Chavarria E, Taura P, Closa D, Boado MA, Ferrer J. Prospective randomized trial of the effect of octreotide on pancreatic juice output after pancreaticoduodenectomy in relation to histological diagnosis, duct size and leakage. HPB (Oxford). 2013 May;15(5):392-9. doi: 10.1111/j.1477-2574.2012.00608.x. Epub 2012 Nov 19. PMID 23557411
- [Result] Yeo CJ, Cameron JL, Lillemoe KD, Sauter PK, Coleman J, Sohn TA, Campbell KA, Choti MA. Does prophylactic octreotide decrease the rates of pancreatic fistula and other complications after pancreaticoduodenectomy? Results of a prospective randomized placebo-controlled trial. Ann Surg. 2000 Sep;232(3):419-29. doi: 10.1097/00000658-200009000-00014. PMID 10973392
- [Result] Montorsi M, Zago M, Mosca F, Capussotti L, Zotti E, Ribotta G, Fegiz G, Fissi S, Roviaro G, Peracchia A, et al. Efficacy of octreotide in the prevention of pancreatic fistula after elective pancreatic resections: a prospective, controlled, randomized clinical trial. Surgery. 1995 Jan;117(1):26-31. doi: 10.1016/s0039-6060(05)80225-9. PMID 7809832